CLINICAL TRIAL: NCT04480697
Title: A Randomized, Double-Blind, Placebo Controlled, Single and Multiple Ascending Doses (SAD/MAD) Study Following Oral Administration in Healthy Subjects to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HPG1860
Brief Title: Study of Safety, Tolerability and PK, PD of HPG1860 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hepagene (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HPG1860-101
Record Dates: First submitted 2020-07-14; First posted 2020-07-21 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part 1 SAD: 6 cohorts Part 2 MAD: 3 cohorts
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- SAD 10mg (Experimental): A single oral dose of 10 mg
  Interventions: Drug: HPG1860
- SAD 20mg (Experimental): A single oral dose of 20 mg. Food effect will also be assessed at the same dose level.
  Interventions: Drug: HPG1860
- SAD 40mg (Experimental): A single oral dose of 40mg
  Interventions: Drug: HPG1860
- SAD 80 mg (Experimental): A single oral dose of 80 mg
  Interventions: Drug: HPG1860
- SAD 120 mg (Experimental): A single oral dose of 120 mg
  Interventions: Drug: HPG1860
- SAD 150 mg (Experimental): A single oral dose of 150 mg
  Interventions: Drug: HPG1860
- MAD 10mg (Experimental): Dose regimen is once daily 10 mg for 14 consecutive days.
  Interventions: Drug: HPG1860
- MAD 30mg (Experimental): Dose regimen is once daily 30 mg for 14 consecutive days.
  Interventions: Drug: HPG1860
- MAD 90 mg (Experimental): Dose regimen is once daily 90mg for 14 consecutive days.
  Interventions: Drug: HPG1860

INTERVENTIONS:
Drug: HPG1860 — 6 subjects randomized to active compound and 2 subjects randomized to placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single and multiple ascending dose Phase 1study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and food effect of HPG1860 orally administered in healthy subjects.

DETAILED DESCRIPTION:
In SAD and MAD studies, all subjects are randomized in a 3:1 ratio. In SAD study , there are 6 cohorts (8 subjects/cohort) with dose levels of 10mg, 20 mg, 40 mg, 80 mg, 120 mg and 150 mg respectively. Blood samples will be collected for safety, PK and PD assessments. After the completion of Cohort 2 (20 mg) in SAD study, following a 7-day washout period, the same 8 subjects will receive another single oral dose of 20 mg HPG1860 after a standard high fat/high calorie breakfast (the fed condition). PK blood samplings will be collected and Cmax and AUC will be used for assessing the food effect. In MAD study, there are 3 cohorts (8 subjects/cohort) with dose levels of 10mg, 30mg and 90 mg, respectively and dosing regimen is once daily for 14 consecutive days. Blood samples will be collected for safety, PK and PD assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18-55 years old (inclusive), male or female
2. Females must be of non-childbearing potential
3. Have a body mass index (BMI) between 18.0 and 32.0 kg/m2 (inclusive) and weigh at least 50 kg at time of Screening

Exclusion Criteria:

1. Clinically significant history of gastrointestinal, cardiovascular, musculoskeletal, endocrine, hematologic, psychiatric, renal, hepatic, bronchopulmonary, neurologic, immunologic, lipid metabolism disorders, or drug hypersensitivity as determined by the Investigator
2. Taken an investigational drug within 3 months or 5 half-live, whichever is longer from the Screening date
3. Any liver function panel analyte (LFT) value > upper limits of normal reference range
4. Positive blood screen for human immunodeficiency virus (HIV), hepatitis B core (IgG and IgM) and surface antigen (HBsAg), Hepatitis A antibody (IgM), hepatitis C antibody (IgG), or hepatitis E (IgG and IgM) at Screening
5. Any condition or finding that in the opinion of the Principal Investigator or designee would put the subject or study conduct at risk if the subject were to participate in the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2019-09-23 (Actual); Primary Completion 2020-11-25 (Actual); Study Completion 2021-08-07 (Actual)

PRIMARY OUTCOMES:
After single ascending doses, number of subjects with treatment-emergent adverse events(TEAEs) in the HPG1860 dose-level cohorts | Day1-8
  To investigate the safety and tolerability of orally administered SAD of HPG1860 by assessment of AEs, vital signs and clinical laboratory findings.
After multiple ascending doses, number of subjects with treatment-emergent adverse events(TEAEs) in the HPG1860 dose-level cohorts | Day1-21
  To investigate the safety and tolerability of orally administered MAD of HPG1860 by assessment of AEs, vital signs and clinical laboratory findings.

SECONDARY OUTCOMES:
Effect of HPG1860 on Blood Concentration of FGF19 and 7-alpha-hydroxy-4-cholesten-3-one (C4) | SAD: Day 1. MAD: Day 1 and Day14
  To assess blood FGF19 and C4 changes vs placebo after orally administered SAD and MAD of HPG1860
Cmax | SAD: up to 48 hours ; MAD: up to 14 days.
  Maximum observed serum concentration
Tmax | SAD: up to 48 hours ; MAD: up to 14 days.
  Time to reach Cmax
AUClast | SAD: up to 48 hours ; MAD: up to 14 days.
  Area under the curve from the time of dosing to the time of the last measurable concentration
AUCinf | SAD: up to 48 hours ; MAD: up to 14 days.
  Area under the curve from the time of dosing extrapolated to infinity
CL | SAD: up to 48 hours; MAD: up to 14 days
  Apparent total body clearance of the drug from plasma
Vd | SAD: up to 48 hours; MAD: up to 14 days
  Apparent volume of distribution
Effect of Food on Cmax of HPG1860 | up to 48 hours
  To assess the effect of food on a single dose of 20 mg HPG1860 by evaluating Cmax
Effect of Food on AUCinf of HPG1860 | up to 48 hours
  To assess the effect of food on a single dose of 20 mg HPG1860 by evaluating AUCinf
Effect of Food on AUC0-24h of HPG1860 | 24 hours
  To assess the effect of food on a single dose of 20 mg HPG1860 by evaluating AUC0-24h

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmaron CPC InC, Baltimore, Maryland, United States